CLINICAL TRIAL: NCT00508196
Title: Endothelial Function and Cardiac Output in Right Ventricular Pacing
Brief Title: Endothelial Function and Cardiac Output in RV Pacing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 190906ver3
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Bradycardia
Keywords: right ventricular pacing; endothelial function; cardiac output
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: RVP-min — DDD pacing with long AV delay
  Other Names: DDD Long
Other: RVP-max — DDD pacing with short AV delay
  Other Names: DDD short

SUMMARY:
Pacing from the right ventricle (as is current practice in patients implanted with permanent pacemakers for bradycardia), has been associated with worse outcomes particularly in heart failure patients. Recent clinical trials suggest that chronic right ventricular pacing (VP) is associated with worsening heart failure, increased strokes and atrial fibrillation. Hemodynamically, right VP results in delayed activation and contraction of the LV which can give rise to functional mitral regurgitation, shortened diastolic filling time and thus reduced coronary filling, as well as abnormal arterial pulsatile flow. The mechanisms for the deleterious effects of right VP in heart failure patients have not been previously investigated. Our aim of this study is therefore to investigate the hemodynamic effects of right VP in stable heart failure patients in terms of exercise cardiac output (CO, an important measure of myocardial function and prognosis), as well as endothelial function which may be deranged as a result of abnormal arterial pulsatile flow.

DETAILED DESCRIPTION:
Study Aims The aim of this study is to investigate the effect of right ventricular pacing on CO at rest and exercise, and on endothelial function and B-type natriuretic peptide, BNP, in patients with heart failure.

Methods: Thirty patients with dual chamber pacemakers for sinus node disease will be recruited: 15 controls with normal LV function and 15 with stable impaired LV function (ejection fraction <40%). The pacemaker will be programmed to pace to back-up pacing at 55bpm in the atrial only (AAI, no right VP) for one week (baseline); and than programmed to overdrive pacing at 70-80bpm, randomised to either to dual chamber, DDD (sequential atrial and ventricular pacing) with a short AV delay (to ensure maximal right VP) or AAI (no RV pacing), for 1 week. There will be a crossover after a 1 week washout at backup AAI pacing at 55 bpm. Resting and exercise CO will be measured at the end of each pacing mode intervention using the Inocor system (a validated non invasive method of CO measurement, using inhaled inert gas equilibriums). Endothelial function will be measured non-invasively at the same time points, as will plasma BNP, a measure of LV strain. Patients with unstable heart failure or angina will be excluded.

Study Endpoints: Rest and exercise CO; and endothelial function and BNP with and without RV pacing, in patients with preserved and impaired LV function.

ELIGIBILITY:
Inclusion Criteria:

* Dual chamber pacemaker
* Intact AV node function

Exclusion Criteria:

* Unstable angina, heart failure
* Inability to exercise

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Struthers, MD, Study Director — University of Dundee
Locations (1):
- Ninewells Hospital and medical School, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects previously implanted with a dual-chamber pacemaker for SND were recruited from the Ninewells Hospital and Medical School pacemaker clinic. No subject was pacemaker dependent and the indication for pacing was intermittent sinus arrest or sinus bradycardia.
Pre-assignment Details: Prior to randomization, as pre-study right ventricular pacing was variable among the subjects, pacing was programmed to produce minimal right ventricular pacing (using single-chamber atrial pacing or dual-chamber mode with long AV delay) for a minimal washout period of ≥1 week.
Groups:
- RVP-Max First, Then RVP-Min: maximum RV pacing programmed (short AV delay) for 1 week, then at least 1 week washout, then minimum RV pacing (long AV delay)
- RVP-Min First, Then RVP-Max: Minimum RV pacing programmed (long AV delay) for 1 week, then at least 1 week washout, then maximum RV pacing (short AV delay)
Period: Overall Study
Arm/Group | RVP-Max First, Then RVP-Min | RVP-Min First, Then RVP-Max
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All subjects had the right ventricular lead implanted at the right ventricular apex. No subject was pacemaker dependent and the indication for pacing was intermittent sinus arrest or sinus bradycardia. Subjects with ongoing angina or heart failure symptoms, known AV node disease, bundle branch block, age >80 years, atrial fibrillation, or inability to exercise, were excluded.
Arm/Group | All Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Function Assessed by Flow Mediated Vasodilatation
Description: Flow mediated vasodilatation as measured by reactive hyperaemia peripheral arterial tonometry signal using EndoPAT software, Itamar.
  A post-occlusion to pre-occlusion ratio is calculated by the EndoPAT software, providing the EndoPAT index (EnFI)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: EndoPAT index (EnFI)
Groups:
- RVP-min: Minimal RV pacing , with long AV delay programmed in DDD mode
- RVP-Max: Maximum RV pacing with short AV delay programmed in DDD mode
Arm/Group | RVP-min | RVP-Max
Number analyzed (Participants) | 22 | 22
EndoPAT index (EnFI) | 1.96 (.37) | 1.73 (0.33)

2. Secondary Outcome: B-type Natriuretic Pepetide
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: microgrammes /L
Arm/Group | RVP-min | RVP-Max
Number analyzed (Participants) | 22 | 22
microgrammes /L | 104.3 (108) | 112.8 (80.2)

3. Secondary Outcome: Cardiac Output
Description: measured at peak exercise on a standard exercise bicycle, measured non-invasively using the inert gas rebreathing technique (Innocor, Innovision A/S, Odense, Denmark).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | RVP-min | RVP-Max
Number analyzed (Participants) | 22 | 22
L/min | 7.65 (3.15) | 7.05 (2.61)

ADVERSE EVENTS:
Arm/Group | RVP-min | RVP-Max
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes